CLINICAL TRIAL: NCT04731246
Title: Video-oculography and Parkinson's Disease: A Prospective Study
Brief Title: Video-oculography and Parkinson's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Association de Recherche Bibliographique pour les Neurosciences (Other)
Collaborators: Centre Hospitalier Princesse Grace (Other); Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: EYE-PD
Record Dates: First submitted 2021-01-20; First posted 2021-01-29 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Parkinson Disease, Idiopathic
Keywords: Parkinson's disease; Video-oculography; Oculomotor disorders; Oculomotricity; Neuropsychological evaluations; Movement disorder; Motor disorders; Non-motor fluctuations
MeSH Terms: conditions — Parkinson Disease; Movement Disorders; Motor Disorders

STUDY DESIGN:
Intervention Model Description: Prospective, descriptive, interventional, monocentric study. Participants perform an annual evaluation, which combine neurological and neuropsychological evaluations and a video-oculography examination.
  Follow-up is carried out over 7 years.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Parkinson's disease (mild to moderate stage) (Experimental)
  Interventions: Other: Video-oculography / Neuropsychological evaluations

INTERVENTIONS:
Other: Video-oculography / Neuropsychological evaluations — Annual evaluation: Medical history; Clinical, Neurological and Neuropsychological evaluations; Video-oculography examination; Inventory of examinations carried out in routine care (brain MRI, cerebral DaTScan, cerebral F-Dopa PET/CT scan, MIBG myocardial scintigraphy, blood test). Follow-up is carried out over 7 years.

SUMMARY:
This study aims to study, in patient with Parkinson's disease, mild to moderate stage (according to Movement Disorder Society Clinical Diagnostic Criteria for Parkinson's Disease, Postuma et al., 2015):

* the evolution of oculomotricity markers over time.
* the correlation between neurological evaluations (motor and non-motor scores), neuropsychological evaluations (cognitive disorders) and oculomotricity evaluation, over a follow-up period of 7 years.
* the impact of antiparkinsonian drugs on the evolution of oculomotricity assessment by video-oculography.
* the value of oculomotricity assessment by video-oculography as an evolutionary marker of the disease.

ELIGIBILITY:
*Inclusion Criteria:

1. Male or Female;
2. Clinically defined idiopathic Parkinson's Disease (PD);
3. Brain MRI performed in routine care in the 12 months preceding inclusion;
4. Cerebral DaTSCAN or cerebral PET with F-DOPA, performed as routine care before inclusion (no time limit), confirming presynaptic dopaminergic denervation;
5. Hoehn & Yahr score: 1 to 3;
6. Normal clinical examination of oculomotricity (slight impairment of smooth pursuit accepted);
7. Neuro-cognitive disorders: absent or minor (according to DSM5);
8. Sufficient written and oral expression in French;
9. Covered by a health insurance system;
10. Written informed consent signed by the patient;
11. Presence of a caregiver.

    * Exclusion Criteria:
12. Psychiatric comorbidity (except anxiety or mild to moderate depression);
13. Neurological comorbidity, if significant;
14. Brain MRI showing:

    1. significant cerebrovascular pathology (Fazekas I admitted),
    2. another brain disease, including stroke.
15. Major cognitive impairment;
16. Absolute exclusion criteria and "Red flags" of the 2015 criteria orienting towards another degenerative pathology of the extrapyramidal system:

    * Cerebellar syndrome
    * Vertical oculomotricity disorders on clinical examination
    * Motor symptoms restricted to the lower limbs
    * Bilateral and perfectly symmetrical parkinsonism
    * Early dystonia
    * Clinical profile suggestive of behavioral variant frontotemporal dementia (bvFTD)
    * Progressive aphasia or apraxia
    * Moderate or severe postural instability and / or early falls
    * Early bulbar dysfunction (dysarthria, swallowing disorders)
    * Ventilatory dysfunction (inspiration)
    * Severe dysautonomia
    * DOPA-resistance
    * Neuroleptic treatment or related
17. Normal MIBG myocardial scintigraphy (if performed).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-07-07 (Actual); Primary Completion 2032-01 (Estimated); Study Completion 2032-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline of Oculomotor raw performance at 7 years - Latency in Horizontal saccades. | Baseline; Year 7
  This concerns saccades Latency (in ms) during horizontal paradigms. Eye movements were recorded and analyzed with an eye-tracking device.
  For each subject value were judged abnormal if they differed by >1.65 SD compared to their reference sample.
Change from Baseline of Oculomotor raw performance at 7 years - Main velocity in Horizontal saccades. | Baseline; Year 7
  This concerns saccades Main velocity (in °/sec) during horizontal paradigms. Eye movements were recorded and analyzed with an eye-tracking device.
  For each subject value were judged abnormal if they differed by >1.65 SD compared to their reference sample.
Change from Baseline of Oculomotor raw performance at 7 years - Gain in Horizontal saccades. | Baseline; Year 7
  This concerns saccades Gain (gaze accuracy) during horizontal paradigms. Eye movements were recorded and analyzed with an eye-tracking device.
  For each subject value were judged abnormal if they differed by >1.65 SD compared to their reference sample.
Change from Baseline of Oculomotor raw performance at 7 years - Latency in Vertical saccades. | Baseline; Year 7
  This concerns saccades Latency (in ms) during vertical paradigms. Eye movements were recorded and analyzed with an eye-tracking device.
  For each subject value were judged abnormal if they differed by >1.65 SD compared to their reference sample.
Change from Baseline of Oculomotor raw performance at 7 years - Main velocity in Vertical saccades. | Baseline; Year 7
  This concerns saccades Main velocity (in °/sec) during vertical paradigms. Eye movements were recorded and analyzed with an eye-tracking device.
  For each subject value were judged abnormal if they differed by >1.65 SD compared to their reference sample.
Change from Baseline of Oculomotor raw performance at 7 years - Gain in Vertical saccades. | Baseline; Year 7
  This concerns saccades Gain (gaze accuracy) during vertical paradigms. Eye movements were recorded and analyzed with an eye-tracking device.
  For each subject value were judged abnormal if they differed by >1.65 SD compared to their reference sample.
Change from Baseline of Inhibition capacity at 7 years | Baseline; Year 7
  Measure of inhibition capacity performance during an "antisaccades" paradigm. Eye movements were recorded and analyzed with an eye-tracking device. Evaluation criteria: percentage of errors. For each subject value were judged abnormal if they differed by >1.65 SD compared to their reference sample.
Change from Baseline of Internuclear ophthalmoplegia (INO) detection at 7 years | Baseline; Year 7
  Highlight presence/absence of INO. Eye movements were recorded and analyzed with an eye-tracking device. Evaluation criteria: INO is present if calculated ratio of abducting to adducting eye movement (both mean and peak velocity) is >1.
Change from Baseline of Fixations impairments detection at 7 years | Baseline; Year 7
  Highlight presence/absence of Fixations impairments. Eye movements were recorded and analyzed with an eye-tracking device. Evaluation criteria: presence/absence/frequency of square wave-jerks, nystagmus, flutters.

SECONDARY OUTCOMES:
Patients description | Baseline
  Profile description of included patients, based on demographic data and clinical exam (sex, age, Weight, height), inclusion/exclusion criteria, medical history, concomitant treatments.
Treatments of Parkinson's disease | Baseline; Year 1; Year 2; Year 3; Year 4; Year 5; Year 6; Year 7: before and after first PD treatment introduction if applicable
  Description of PD treatments of included patients (Name, start date, end date, dose).
Evolution of Oculomotor raw performance - Latency in Horizontal saccades | Baseline; Year 1; Year 2; Year 3; Year 4; Year 5; Year 6; Year 7: before and after first PD treatment introduction if applicable
  This concerns saccades Latency (in ms) during horizontal paradigms. Eye movements were recorded and analyzed with an eye-tracking device.
  For each subject value were judged abnormal if they differed by >1.65 SD compared to their reference sample. Parameter used for description, evolution and correlation studies.
Evolution of Oculomotor raw performance - Main velocity in Horizontal saccades. | Baseline; Year 1; Year 2; Year 3; Year 4; Year 5; Year 6; Year 7: before and after first PD treatment introduction if applicable
  This concerns saccades Main velocity (in °/sec) during horizontal paradigms. Eye movements were recorded and analyzed with an eye-tracking device.
  For each subject value were judged abnormal if they differed by >1.65 SD compared to their reference sample. Parameter used for description, evolution and correlation studies.
Evolution of Oculomotor raw performance - Gain in Horizontal saccades. | Baseline; Year 1; Year 2; Year 3; Year 4; Year 5; Year 6; Year 7: before and after first PD treatment introduction if applicable
  This concerns saccades Gain (gaze accuracy) during horizontal paradigms. Eye movements were recorded and analyzed with an eye-tracking device.
  For each subject value were judged abnormal if they differed by >1.65 SD compared to their reference sample. Parameter used for description, evolution and correlation studies.
Evolution of Oculomotor raw performance - Latency in Vertical saccades | Baseline; Year 1; Year 2; Year 3; Year 4; Year 5; Year 6; Year 7: before and after first PD treatment introduction if applicable
  This concerns saccades Latency (in ms) during vertical paradigms. Eye movements were recorded and analyzed with an eye-tracking device.
  For each subject value were judged abnormal if they differed by >1.65 SD compared to their reference sample. Parameter used for description, evolution and correlation studies.
Evolution of Oculomotor raw performance - Main velocity in Vertical saccades | Baseline; Year 1; Year 2; Year 3; Year 4; Year 5; Year 6; Year 7: before and after first PD treatment introduction if applicable
  This concerns saccades Main velocity (in °/sec) during vertical paradigms. Eye movements were recorded and analyzed with an eye-tracking device.
  For each subject value were judged abnormal if they differed by >1.65 SD compared to their reference sample. Parameter used for description, evolution and correlation studies.
Evolution of Oculomotor raw performance - Gain in Vertical saccades | Baseline; Year 1; Year 2; Year 3; Year 4; Year 5; Year 6; Year 7: before and after first PD treatment introduction if applicable
  This concerns saccades Gain (gaze accuracy) during vertical paradigms. Eye movements were recorded and analyzed with an eye-tracking device.
  For each subject value were judged abnormal if they differed by >1.65 SD compared to their reference sample. Parameter used for description, evolution and correlation studies.
Inhibition capacity | Baseline; Year 1; Year 2; Year 3; Year 4; Year 5; Year 6; Year 7: before and after first PD treatment introduction if applicable
  Measure of inhibition capacity performance during an "antisaccades" paradigm. Eye movements were recorded and analyzed with an eye-tracking device. Evaluation criteria: percentage of errors. For each subject value were judged abnormal if they differed by >1.65 SD compared to their reference sample. Parameter used for description, evolution and correlation studies.
Internuclear ophthalmoplegia (INO) detection | Baseline; Year 1; Year 2; Year 3; Year 4; Year 5; Year 6; Year 7: before and after first PD treatment introduction if applicable
  Highlight presence/absence of INO. Eye movements were recorded and analyzed with an eye-tracking device. Evaluation criteria: INO is present if calculated ratio of abducting to adducting eye movement (both mean and peak velocity) is >1. Parameter used for description, evolution and correlation studies.
Fixations impairments detection | Baseline; Year 1; Year 2; Year 3; Year 4; Year 5; Year 6; Year 7: before and after first PD treatment introduction if applicable
  Highlight presence/absence of Fixations impairments. Eye movements were recorded and analyzed with an eye-tracking device. Evaluation criteria: presence/absence/frequency of square wave-jerks, nystagmus, flutters. Parameter used for description, evolution and correlation studies.
Neurological evaluation - evolution of motor disorders | Baseline; Year 1; Year 2; Year 3; Year 4; Year 5; Year 6; Year 7: before and after first PD treatment introduction if applicable
  Motor disorders are applause sign, Pyramidal signs, conjugate oculomotricity disorders, cerebellar syndrome. They are categorised as present/absent following neurological clinic evaluation. These parameters are used for description, evolution and correlation analysis.
Neurological evaluation - Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III | Baseline; Year 1; Year 2; Year 3; Year 4; Year 5; Year 6; Year 7: before and after first PD treatment introduction if applicable
  Score on the Part III subscale of the MDS-UPDRS, that assesses the motor signs of PD. Scores range from 0-33 with a lower score indicating less severe impairment. These scores are used for description, evolution and correlation studies.
Neurological evaluation - Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part IV | Baseline; Year 1; Year 2; Year 3; Year 4; Year 5; Year 6; Year 7: before and after first PD treatment introduction if applicable
  Score on the Part IV subscale of the MDS-UPDRS, that assesses the motor complications of PD. Scores range from 0-6 with a lower score indicating less severe impairment. These scores are used for description, evolution and correlation studies.
Neurological evaluation - Movement Disorder Society Non-Motor rating Scale (MDS-NMS) | Baseline; Year 1; Year 2; Year 3; Year 4; Year 5; Year 6; Year 7: before and after first PD treatment introduction if applicable
  This Non-Motor rating Scale measures frequency and severity of 13 non-motor domains, over 52 items, and covers a range of key non-motor symptoms both PD and treatment related. The MDS-NMS total score is the sum of the 13 non-motors domains subscales scores (these subscales' scores are the sum of the frequency multiplied by the intensity of each items composing each 13 non-motor domains). Higher score means a worse outcome. Score range 0-832. These scores are used for description, evolution and correlation studies.
Neurological evaluation - Movement Disorder Society Non-Motor rating Scale (MDS-NMS) Non-Motor Fluctuations (NMF) | Baseline; Year 1; Year 2; Year 3; Year 4; Year 5; Year 6; Year 7: before and after first PD treatment introduction if applicable
  The MDS-NMS has a Non-Motor Fluctuations subscale (NMF) to assess changes in non-motor symptoms in relation to the timing of anti-parkinsonian medications across 8 domains. The MDS-NMS NMF Total score is the Subscore "Change" (range 0-32) multiplied by Subscore "Time" (range 1-4). The MDS-NMS NMF Total score range is 0-128. Higher score means a worse outcome.
  This score is used for description, evolution and correlation studies. [Time Frame: Baseline; Year 1; Year 2; Year 3; Year 4; Year 5; Year 6; Year 7: before and after first PD treatment introduction if applicable]
Orthostatic hypotension | Baseline; Year 1; Year 2; Year 3; Year 4; Year 5; Year 6; Year 7: before and after first PD treatment introduction if applicable
  Blood pressure measures in order to determine presence or absence of Orthostatic hypotension. These parameters are used for description, evolution and correlation studies.
MRI scan | Baseline; Year 3; Year 7
  Brain MRI data described according to their nature (lesion / atrophy / anomaly / Score Fasekas) are classified as normal or abnormal.
DAT scan | Baseline; Year 3; Year 7
  Cerebral DAT-Scan data are classified as presence/absence of Dopaminergic denervation.
PET/CT scan | Baseline; Year 3; Year 7
  Cerebral F-Dopa PET/CT-Scan data are classified as presence/absence of Dopaminergic denervation.
MIBG myocardial scintigraphy | Baseline; Year 3; Year 7
  MIBG myocardial scintigraphy are classified as normal/abnormal.
Mini Mental State (MMSE) | Baseline; Year 1; Year 2; Year 3; Year 4; Year 5; Year 6; Year 7
  Mini Mental State (MMSE) is used to evaluate Global cognitive performance. MMSE is a 30-question general cognitive function assessment. The maximum score is 30. Performance of each participant is compared to their reference sample (depending on age, sex and level study). Scores are used for description, evolution and correlation studies.
Evolution of general cognitive behavior | Baseline; Year 1; Year 2; Year 3; Year 4; Year 5; Year 6; Year 7
  The Mattis Dementia Rating Scale is used to to evaluate general cognitive behavior of subjects with suspected dementia. The scale is made up of 36 items divided into 5 complementary parts, each corresponding to a cognitive function: attention, initiation, construction, conceptualization, memory. The total score is /144 points. Score is used for description, evolution and comparison studies. Higher score means a better outcome.
Episodic memory performance | Baseline; Year 1; Year 2; Year 3; Year 4; Year 5; Year 6; Year 7
  The GROBER et BUSCHKE Free and Cued recall (16 items) is used to evaluate Episodic memory. Performances of each participant are compared to their reference sample (depending on age, sex and level study). These parameters are used for description, evolution and correlation studies.
Executive performance - T.M.T | Baseline; Year 1; Year 2; Year 3; Year 4; Year 5; Year 6; Year 7
  Trail Making Test (T.M.T) A&B is used to evaluate executive performance. The task requires a subject to connect a sequence of 25 consecutive targets on a sheet of paper, in the shortest time possible without lifting the pen from the paper. Time performances of each participant are compared to their reference sample. These parameters are used for description, evolution and correlation studies.
Executive performance - Stroop test | Baseline; Year 1; Year 2; Year 3; Year 4; Year 5; Year 6; Year 7
  Stroop test (GREFFEX) is used to evaluate executive performance and more specifically inhibition. The time to complete each condition (in seconds) is recorded, as well as the number of uncorrected and corrected errors. Stroop task performances of each participant are compared to their reference sample. These parameters are used for description, evolution and correlation studies.
Executive performance - B.R.E.F. | Baseline; Year 1; Year 2; Year 3; Year 4; Year 5; Year 6; Year 7
  The "Batterie rapide d'évaluation frontale" (B.R.E.F.), or Frontal Assessment Battery at Bedside (F.A.B.), is used to determine the presence or not of a cognitive and behavioral dysexecution syndrom. The maximum score is 18. Performances of each participant are compared to their reference sample. These parameters are used for description, evolution and correlation studies.
Verbal fluency | Baseline; Year 1; Year 2; Year 3; Year 4; Year 5; Year 6; Year 7
  Verbal fluency test is a short test of verbal functioning. It consists of two tasks: category fluency and letter fluency. Participant is given 1 minute to produce as many unique words as possible within a semantic category (category fluency) or starting with a given letter (letter fluency). The participant's score in each task is the number of unique correct words. Performances of each participant are compared to their reference sample. These parameters are used for description, evolution and correlation studies.
Visuospatial function | Baseline; Year 1; Year 2; Year 3; Year 4; Year 5; Year 6; Year 7
  Visual Object and Space Perception battery (VOSP) consists of eight tests each designed to assess a particular aspect of object or space perception, while minimizing the involvement of other cognitive skills. Performance of each participant is compared to their reference sample.
  This parameter is used for description, evolution and comparison studies.
Visuospatial/constructional ability | Baseline; Year 1; Year 2; Year 3; Year 4; Year 5; Year 6; Year 7
  Rey-complex copy figure test is used to evaluate visuospatial/constructional abilities. Performance of each participant is compared to their reference sample. These parameters are used for description, evolution and comparison studies.
Praxis assessment | Baseline; Year 1; Year 2; Year 3; Year 4; Year 5; Year 6; Year 7
  Praxies idéomotrices (Mahieux) is a neuropsychological measure of imitation of meaningless gestures (score /8), symbolic gestures (score /5), pantomimes (score /10). Motor praxis are also measured (kinesthetic praxis, melokinetic praxis). These parameters are used for description, evolution and correlation analysis.
Social cognition and Emotional assessment | Baseline; Year 1; Year 2; Year 3; Year 4; Year 5; Year 6; Year 7
  A test battery made up of the Faux pas recognition test and a facial emotion recognition test (The Mini-sea) are used to evaluate Social cognition and Emotional assessment.
  Evaluation criteria: Score to The Faux pas recognition test (/15), and scores to facial emotion recognition test (total score / 35 and sub-scores / 5). Performances of each participant are compared to their reference sample.
  These parameters are used for description, evolution and correlation studies.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe BARRES, MD, Study Director — Centre Mémoire, Centre de Gérontologie Clinique RAINIER III, Princess Grace Hospital, Monaco.; Sandrine LOUCHART DE LA CHAPELLE, MD-PHD, Principal Investigator — Centre Mémoire, Centre de Gérontologie Clinique RAINIER III, Princess Grace Hospital, Monaco; Alain PESCE, PUPH, Study Chair — AREBISN (Association de Recherche Bibliographique pour les Neurosciences), Nice (France); Caroline GIORDANA, MD, Principal Investigator — Centre Expert Parkinson, Unités des Pathologies du Mouvement, Hôpital Pasteur 2, Nice (France); Benoit PAULMIER, MD, Principal Investigator — Médecine Nucléaire, Princess Grace Hospital, Monaco.
Locations (1):
- Centre Mémoire / Centre de Gérontologie Clinique Rainier III / Princess Grace Hospital, Monaco, Monaco

IPD SHARING:
Plan to Share IPD: No